CLINICAL TRIAL: NCT06870383
Title: Analgesic Efficacy of Erector Spinae Plane Block Versus Combined Pecto-intercostal and Recto-intercostal Fascial Plane Block in Patients Undergoing Cardiac Surgery: A Randomized Comparative Trial
Brief Title: Erector Spinae Block Versus Combined Pecto-intercostal and Recto-intercostal Fascial Plane Block in Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, lecturer of anesthesiology, surgical intensive care and pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR1085/2/25
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Erector Spinae Plane Block; Pecto-intercostal Fascial Plane Block; Recto-intercostal Fascial Plane Block; Cardiac; Surgery
Keywords: Analgesic; Erector; Pectointercostal; Rectointercostal; Cardiac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (Active Comparator): At the level of fourth thoracic vertebra, the ultrasound transducer (5-14 Mhz) Philips CX50 will be placed in the sagittal plane and moved 3 cm to visualize the transverse process of T4 or T5 with erector spinae muscle overlying it, the needle will be inserted in plane into the facial plane deep to the erector spinae muscle with the tip contacting the transverse process of T4 or T5. After confirmation by 5 ml saline, 20 ml bupivacaine 0.25% will be injected for each side ensuring not to exceed the maximal 2 mg/kg bupivacaine dose.
  Interventions: Drug: Erector spinae plane block
- Combined Pecto-intercostal and recto-intercostal fascial plane block group (Experimental): A high-frequency ultrasound transducer will be placed 2 cm lateral to sternal edge at the level of 4th rib. A needle will be inserted in-plane under ultrasound guidance through the pectoralis major muscle, and the drug will be deposited in the pecto-intercostal fascial plane located between the pectoralis major muscle and the fourth rib (or intercostal muscle) after confirmation by 5 ml saline. 10-15 mL of 0.25% bupivacaine will be injected for each side. Then the transducer will be placed 2-3 cm lateral and caudal to the xiphoid in the epigastric area.The needle will be inserted between RAM and the costal cartilages with an in-plane technique in a caudo-cranial way. Hydro-dissection will be performed with 5 ml saline for confirmation needle tip position, 10-15 mL of 0.25% bupivacaine will be injected for each side.
  Interventions: Drug: Combined Pecto-intercostal and recto-intercostal fascial plane block

INTERVENTIONS:
Drug: Erector spinae plane block — The block will be done under ultrasound guidance using 20 ml bupivacaine 0.25% that will be injected for each side ensuring not to exceed the maximal 2 mg/kg bupivacaine dose.
  Arms: Erector spinae plane block group
Drug: Combined Pecto-intercostal and recto-intercostal fascial plane block — The blocks will be done under ultrasound guidance using 10-15 ml of 0.25% bupivacaine that will be injected for each side ensuring not to exceed the maximal 2 mg/kg bupivacaine dose..
  Arms: Combined Pecto-intercostal and recto-intercostal fascial plane block group

SUMMARY:
The aim of this study is to compare the analgesic effects of ultrasound-guided bilateral erector spinae plane block versus ultrasound-guided bilateral combined Pecto-intercostal fascial plane block and recto-intercostal fascial plane block in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
The incidence of severe acute postoperative pain after median sternotomy is as high as 49 %. A number of regional techniques have been used to treat sternotomy pain such as thoracic epidural, intercostal nerve block, paravertebral nerve block & thoracic erector spinae plane block which has been used extensively in cardiac surgery providing adequate postoperative pain control. Pecto-intercostal fascial plane block is a minimally invasive, regional fascial plane block technique that can be administered as a part of a multimodal analgesic regimen. It targets the anterior intercostal nerves as they run in the fascial plane between the pectoralis major muscle and the external intercostal muscles and emerge on either side of the sternum. Recently, Tulgar et al. have described a novel block named "recto-intercostal fascial plane block" which is performed between the rectus abdominis muscle and costal cartilages of ribs 6-7 (insertion of RAM). In their cadaveric examination, they reported that the dye spread extensively to the anterior branches of the T6-T9 thoracic nerves, and laterally to the entire lower thorax. The investigators assume that the incomplete dermatome coverage by Pecto-intercostal fascial plane block might be responsible for its inferior analgesic quality compared to erector spinae plane block which was reported in some previous reports. So, the investigators will conduct this novel study to investigate and compare the analgesic effects of erector spinae plane block and combined Pecto-intercostal fascial plane block and recto-intercostal fascial plane block in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 65 years.
* Both sexes.
* Scheduled for open heart surgery with cardiopulmonary bypass and midline sternotomy.

Exclusion Criteria:

* History of chronic pain or Long-term or recent use of opioids.
* History of allergy to local anesthetic drugs.
* Ejection fraction of left ventricle less than 30%.
* History of psychiatric diseases or any neurological disorders.
* Pre-existing major organ dysfunction as hepatic or renal failure.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
The total opioid consumption in first 24 hours after surgery. | 24 hours after surgery.
  opioid analgesia will be given if the pain scores ≥ 4.

SECONDARY OUTCOMES:
Intraoperative fentanyl dose | Until the end of surgical procedure.
  Fentanyl bolus dosages of 2μg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline.
Postoperative pain scores after extubation, at 8, 12, 18, 24, 36, and 48 hour after surgery. | 48 hours after surgery.
  Numerical rating scale pain score (NRS) ranges from 0= no pain to 10= worst pain will be used to evaluate pain scores after surgery.
Extubation time | 24 hours after surgery.
  Time from intensive care unit admission until successful removal of endotracheal tube will be recorded.
Side effects | 24 hours after surgery.
  Hypotension , bradycardia, postoperative nausea and vomiting
Incidence of chronic pain at 3, and 6 months after surgery. | 6 months after surgery.
  chronic pain will be assessed and its severity graded by rating scale will be recorded.
Opioid consumption in the second day after surgery. | 48 hours after surgery.
  opioid analgesia will be given if the pain scores ≥ 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the study.
Access Criteria: The data will be available upon reasonable request from the corresponding author.